CLINICAL TRIAL: NCT01542801
Title: Comparison of Daily Norfloxacin Versus Weekly Ciprofloxacin for the Prevention of Spontaneous Bacterial Peritonitis in Cirrhotic Patients
Brief Title: Norfloxacin Versus Ciprofloxacin for Spontaneous Bacterial Peritonitis (SBP) Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: Sungkyunkwan University (Other); Kyungpook National University Hospital (Other); Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Soon Ho Um, Professor of Medicine, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBP_prevention
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Adverse Reaction to Other Drugs and Medicines
Keywords: Effect of Preventive Antibiotics
MeSH Terms: interventions — Norfloxacin; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norfloxacin (Active Comparator): norfloxacin 400 mg once daily administration
  Interventions: Drug: Norfloxacin
- Ciprofloxacin (Experimental): Ciprofloxacin 750 mg per week
  Interventions: Drug: ciprofloxacin

INTERVENTIONS:
Drug: Norfloxacin — Norfloxacin 400 mg per day
  Arms: Norfloxacin
Drug: ciprofloxacin — Ciprofloxacin 750 mg per week
  Arms: Ciprofloxacin

SUMMARY:
* For the prevention of spontaneous bacterial peritonitis (SBP) in patients with liver cirrhosis, norfloxacin 400mg per day is a standard regimen.
* Ciprofloxacin 750 mg per week is also known to be effective for prevention of SBP. In addition, ciprofloxacin once weekly administration is more convenient and less costly.
* Therefore ciprofloxacin once weekly could be more useful if the the efficacy is comparable to norfloxacin once daily.
* This study aims to prove ciprofloxacin once weekly administration is as effective as norfloxacin once daily administration for the prevention of SBP in cirrhotic patients with ascites.

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP) is one of the most serious complication of liver cirrhosis.

The short term mortality reaches 20-30% mainly due to sepsis, hepatorenal syndrome, and liver failure. In addition, patients who suffered SBP show poor prognosis with 1 year-mortality of 50-70%. The high recurrence rate is also problematic. Therefore appropriate prevention of SBP is critically needed to improve survival as well as quality of life.

Selective intestinal decontamination (SID) is eradicating gram negative bacterial in the gut lumen, and effectively prevent development of SBP. Patients with gastrointestinal hemorrhage, low ascitic protein level, high bilirubin, or history of SBP need SID.

Norfloxacin 400 mg daily administration decreased the incidence of SBP to 2% compared with 17% of no prevention group's among patients with ascitic protein less than 1.5 g/dL. Also, in high risk patients (Child-Pugh score > or = 9 points and serum bilirubin level > or = 3 mg/dL, serum creatinine level > or = 1.2 mg/dL, blood urea nitrogen level > or = 25 mg/dL, or serum sodium level < or = 130 mEq/L), norfloxacin 400 mg/day improved 1 year-survival to 60% compared with 48% of no prevention group's. Therefore norfloxacin is now primarily recommend for the prevention of SBP in cirrhotic patients. However, norfloxacin should be administered on daily basis, so efforts to reduce cost and frequency have been made.

Ciprofloxacin 750 mg weekly administration has been evaluated, and shown to be effective as 3.6% versus 22% in prevention versus no prevention arm, respectively. Therefore, ciprofloxacin 750 mg/week is a reasonable option for prevention of SBP. However, comparison of efficacy of these two methods (norfloxacin 400 mg daily versus ciprofloxacin 750 mg weekly) has not been performed, yet.

The investigators aim to compare the efficacy and safety of norfloxacin 400 mg daily and ciprofloxacin 750 mg weekly for the proper management of cirrhotic patients with ascites.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-75 years old
* Liver cirrhosis with ascites
* Ascitic polymorphonucleated cells (PMN) count < 250/mm3
* Ascitic protein <= 1.5 g/dL or History of SBP

Exclusion Criteria:

* Incompatibility with inclusion criteria
* Hypersensitivity or intolerability with quinolones
* Hepatocellular carcinoma beyond Milan Criteria
* Hepatic encephalopathy over stage 2
* History of treatment with antibiotics within 2 weeks of enrollment
* HIV infection
* Untreated malignancy
* Women with child-bearing age not willing to use effective contraception.
* Pregnant or breast feeding women
* Not able to give informed consents

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-08; Primary Completion 2015-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The prevention rate of spontaneous bacterial peritonitis (SBP) | 12 months
  The incidence of SBP will measured in each the group. Thereby, prevention rate will also be compared between the groups.

SECONDARY OUTCOMES:
1 year mortality | 12 months ( 1 year)
  liver related mortality and overall mortality will be assessed.
Incidence of infectious event other than SBP | 12 months
  Bacteremia, urinary tract infection, pneumonia, and other infections will be included.
Hepatorenal syndrome | 12 months
  Diagnostic criteria of hepatorenal syndrome is defined by the latest version of Internation ascites club consensus.
Hepatic encephalopathy | 12 months
  Will follow the Western Heaven Criteria.
Adverse event of drugs | 12 months
  Any of adverse event suspected by study drugs will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Soon Ho Um, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital; Hyung Joon Yim, M.D., Ph.D., Study Director — Korea University Ansan Hospital
Locations (7):
- South Korea (7):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Soonchunhyang University College of Medicine, Bucheon Hospital, Bucheon-si
  - Soonchunhyang University College of Medicine, Cheonan Hospital, Cheonan
  - Kyungpuk National University Hospital, Daegu
  - Korea University Anam Hospital, Seoul
  - Soonchunhyang University College of Medicine, Seoul Hospital, Seoul
  - Sungkyunkwan University Gangbuk Samsung Hospital, Seoul

REFERENCES:
- [Background] Mowat C, Stanley AJ. Review article: spontaneous bacterial peritonitis--diagnosis, treatment and prevention. Aliment Pharmacol Ther. 2001 Dec;15(12):1851-9. doi: 10.1046/j.1365-2036.2001.01116.x. PMID 11736714
- [Background] Koulaouzidis A, Bhat S, Karagiannidis A, Tan WC, Linaker BD. Spontaneous bacterial peritonitis. Postgrad Med J. 2007 Jun;83(980):379-83. doi: 10.1136/pgmj.2006.056168. PMID 17551068
- [Background] Fernandez J, Navasa M, Gomez J, Colmenero J, Vila J, Arroyo V, Rodes J. Bacterial infections in cirrhosis: epidemiological changes with invasive procedures and norfloxacin prophylaxis. Hepatology. 2002 Jan;35(1):140-8. doi: 10.1053/jhep.2002.30082. PMID 11786970
- [Background] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Result] Rolachon A, Cordier L, Bacq Y, Nousbaum JB, Franza A, Paris JC, Fratte S, Bohn B, Kitmacher P, Stahl JP, et al. Ciprofloxacin and long-term prevention of spontaneous bacterial peritonitis: results of a prospective controlled trial. Hepatology. 1995 Oct;22(4 Pt 1):1171-4. doi: 10.1016/0270-9139(95)90626-6. PMID 7557868
- [Result] Grange JD, Roulot D, Pelletier G, Pariente EA, Denis J, Ink O, Blanc P, Richardet JP, Vinel JP, Delisle F, Fischer D, Flahault A, Amiot X. Norfloxacin primary prophylaxis of bacterial infections in cirrhotic patients with ascites: a double-blind randomized trial. J Hepatol. 1998 Sep;29(3):430-6. doi: 10.1016/s0168-8278(98)80061-5. PMID 9764990
- [Result] Fernandez J, Navasa M, Planas R, Montoliu S, Monfort D, Soriano G, Vila C, Pardo A, Quintero E, Vargas V, Such J, Gines P, Arroyo V. Primary prophylaxis of spontaneous bacterial peritonitis delays hepatorenal syndrome and improves survival in cirrhosis. Gastroenterology. 2007 Sep;133(3):818-24. doi: 10.1053/j.gastro.2007.06.065. Epub 2007 Jul 3. PMID 17854593
- See also: Korea University (PI of SBP_prevention study is belong to this university) — http://www.korea.ac.kr